CLINICAL TRIAL: NCT03165825
Title: Pragmatic Randomized Prospective Study of Cervical Interlaminar Epidural Injection of Particulate Steroid and Cervical Transforaminal Epidural Injection of Non-particulate Steroid in Patients With Cervical Radicular Pain
Brief Title: Cervical Interlaminar Versus Transforaminal Epidural Steroid Injection
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: funding
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Byron Schneider, Assistant Professor, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB #170187
Record Dates: First submitted 2017-05-16; First posted 2017-05-24 (Actual); Last update posted 2018-10-04 (Actual); Status verified 2018-10

CONDITIONS: Cervical Radiculopathy
MeSH Terms: conditions — Radiculopathy | interventions — Dexamethasone; Calcium Dobesilate; Betamethasone

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tranforaminal (Experimental): will receive cervical epidural injection via a transforaminal route with dexamethasone steroid
  Interventions: Drug: Transforaminal Epidural Steroid Injection with Dexamethasone
- Interlaminar (Active Comparator): will receive cervical epidural injection via an interlaminar route with betamethasone steroid
  Interventions: Drug: Interlaminar Epidural Steroid Injection with Betamethasone

INTERVENTIONS:
Drug: Transforaminal Epidural Steroid Injection with Dexamethasone — Transforaminal Epidural Steroid Injection with Dexamethasone
  Other Names: Decadron
  Arms: Tranforaminal
Drug: Interlaminar Epidural Steroid Injection with Betamethasone — Interlaminar Epidural Steroid Injection with Betamethasone
  Arms: Interlaminar

SUMMARY:
compare cervical interlaminar epidural injection of betamethasone (9mg) and cervical transforaminal epidural injection of dexamethasone (15 mg) for cervical radicular pain

DETAILED DESCRIPTION:
This study will compare one route of epidural steroid injection (interlaminar) using a particulate steroid to another route of epidural steroid injection (transforaminal) using a different non-particulate steroid dexamethasone. Repeat injections may be allowed.

All injections will be done with image guidance. Patients will be evaluated for improvements in pain and function.

ELIGIBILITY:
Inclusion Criteria:

* - aged >18, capable of understanding and providing consent in English, capable of complying with the outcome instruments used, capable of attending all planned follow up visits
* unilateral cervical radicular pain as defined by arm pain or shoulder girdle pain/periscapular pain with or without neck pain of at least 2 weeks.
* 7 day average of numeric pain rating score (NPRS) for arm pain or shoulder girdle/periscapular pain of at least 5/10 at baseline evaluation
* MRI (or CT if MRI not available) shows one or two level cervical disc herniation(s) or disc osteophyte complex(es) between levels C4-T1, corresponding in location with unilateral radicular pain, with or without neurological deficits. MRI or CT may show degenerative changes at other levels.
* Patient consents to treatment with epidural injection in a shared decision-making process with the treating physician.
* Pain duration of at least 2 weeks or more.

Exclusion Criteria:

* - Neck pain is greater than arm pain or shoulder girdle/periscapular pain based on 7 day average NPRS
* Those receiving remuneration for their pain treatment (e.g., disability, worker's compensation).
* Those involved in active litigation relevant to their pain.
* Those unable to read English and complete the assessment instruments.
* Those unable to attend follow up appointments
* The patient is incarcerated.
* Spondylolisthesis at the involved or adjacent segments.
* History of prior cervical surgery
* Progressive motor deficit, and/or clinical signs of myelopathy.
* Prior cervical epidural steroid injections.
* Prior epidural steroid injection within the prior 12 months in any location within the spine.
* Possible pregnancy or other reason that precludes the use of fluoroscopy.
* Allergy to contrast media or local anesthetics.
* BMI>35.
* Systemic inflammatory arthritis (e.g., rheumatoid arthritis, ankylosing spondylitis, lupus).
* Active infection or treatment of infection with antibiotics within the past 7 days.
* Medical conditions causing significant functional disability (e.g., stroke, COPD)
* Chronic widespread pain or somatoform disorder (e.g. fibromyalgia).
* Addictive behavior, severe clinical depression, or psychotic features.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-01 (Estimated); Primary Completion 2019-09 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
Pain | 12 months
  Numeric rating pain score

CONTACTS AND LOCATIONS:
Overall Officials: Byron Schneider, Principal Investigator — Assistant professor

IPD SHARING:
Plan to Share IPD: No